CLINICAL TRIAL: NCT04166240
Title: Measuring and Improving the Safety of Test Result Follow-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other); Birmingham VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 17-127; H-45450 (Other: Baylor College of Medicine)
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Breast Cancer; Colon Cancer; Bladder Cancer; Hepatocellular Cancer
Keywords: Diagnostic Errors; Quality Improvement; Patient Safety; Delayed Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Urinary Bladder Neoplasms; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: It's a cluster randomized control trial where 12 sites are randomized in groups of 4 in 3 clusters each.
Masking Description: VBTS participants, providers, and outcome assessors know about the intervention and in which conditions sites are in and when.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAFER TRACKS Intervention (Experimental): Each cluster starts receiving the intervention in sequence per cluster randomized control trial designs. Each cluster will participate in attending monthly coaching calls and compare their data on test results from pre-intervention to receiving the intervention.
  Interventions: Behavioral: SAFER TRACKS Intervention
- Non-intervention period (No Intervention): When the cluster is not in active intervention, they are in the non-intervention period. The amount of time that each site contributes to the intervention depends on which cluster they belong to.

INTERVENTIONS:
Behavioral: SAFER TRACKS Intervention — SAFER Change Package delivered using a Virtual Breakthrough Series [VBTS] Collaborative supplemented with automated surveillance data on test results.
  Arms: SAFER TRACKS Intervention

SUMMARY:
Improving communication is foundational to improving patient safety. Electronic health records (EHRs) can improve communication, but also introduce unique vulnerabilities. Failure to follow-up abnormal test results (missed results) is a key preventable factor in diagnosis and treatment delays in the Veteran's Health Administration (VHA) and often involves EHR-based communication breakdowns. Effective methods are needed to detect diagnostic delays and intervene appropriately. Manual techniques to detect care delays, such as spontaneous reporting and random chart reviews, have limited effectiveness, due in part to bias and lack of provider awareness of delays. They are also inefficient and cost-prohibitive when applied to large numbers of patients.

Diagnostic errors are considered harder to tackle, in part because they are difficult to measure. Rigorous measurement of diagnostic safety is essential and should be prioritized given the increasing amount of electronically available data. To create an effective measurement and learning program researchers must (1) ensure teams know how to take actionable steps on data and have assistance in doing so and (2) prioritize diagnostic safety at the organizational level by securing commitment from local VA leadership and clinical operations personnel. This will ensure that safety measurement will translate into action. The proposed study focuses on creating a novel program to develop and evaluate multifaceted socio-technical tools and strategies to help prevent, detect, mitigate, and ameliorate breakdowns in EHR-based communication that often lead to "missed" test results in the VHA.

DETAILED DESCRIPTION:
The goal of this study is to develop and evaluate a new program for surveillance and improvement of test results-related diagnostic safety. The investigators will use a multifaceted measurement approach, the Virtual Breakthrough Series (VBTS) model, to account for processes of care and work systems issues as well as outcomes and implement change.

This is for Aim 2 of the study which was approved under Institutional Review Board (IRB) Protocol Number: H-45450. This study will implement the Change Package which was developed in the research team's recent work (Aim1, prior IRB Protocol Number: H-43661 from October 2018 - September 2019) via Virtual Breakthrough Series using a stepped-wedge cluster-randomized control trial. The study design involves random and sequential crossover of clusters from control to intervention until all clusters are exposed. A Change Package is a catalogue of evidence-based practices, change concepts, and action steps/strategies that help guide improvement efforts. VBTS involves monthly learning sessions where participants are provided with education/review of a specific component of a Change Package along with reviewing de-identified data, and having a facilitated discussion about successes, challenges, and implementation progress related to needed changes. The intervention will consist of coached implementation of the SAFER Change Package using a VBTS Collaborative, plus automated near real-time surveillance data on potentially missed test results through monthly data extraction within the Corporate Data Warehouse (CDW) platform.

The study's outcome measures will be the rate of missed test results, determined through random manual medical record review conducted nationally as part of the VHA performance-measurement system, known as the External Peer Review Program (EPRP) which has been collecting facility-level data on timeliness of communication of test results to patients within the time periods specified by VHA Directive 1088, as well as automated indicators (Triggers) of missed test results. Electronic surveillance will be made possible through the use of the research team's trigger algorithms which will determine the number of patients potentially lost to follow-up for the specified condition based on a previously validated timeframe. The triggers use the national EHR data warehouse (VINCI/CDW) to identify patients at risk for delays or patients who may have fallen through the cracks. For data surveillance, the investigators will apply five triggers to the medical record data contained within the CDW for the participating facilities during the Intervention Phase along with evaluating EPRP data. The research team hypothesizes there will be fewer missed test results in participating sites during the SAFER TRACKS Intervention as compared to during the pre-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Medical records identified via CDW which fall under the EPRP measures (Fecal Occult Blood Test FOBT)/Fecal Immunohistochemical Test (FIT), Hepatitis C Virus (HCV), Mammogram, alpha feto protein (AFP), dual energy x-ray absorptiometry (DEXA) Scan, Pap/ human papillomavirus (HPV), Chest X-ray, and Chest CT)
* Medical records containing clinical findings suspicious for breast cancer, lung cancer, bladder cancer, hepatocellular carcinoma, and colorectal cancer (CRC)

Exclusion Criteria:

* Medical records that don't contain any tests, procedures, or appointments that need to be followed up on

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hardeep Singh, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (2):
- United States (2):
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No
No plans to share individual site data.

REFERENCES:
- [Background] Walter FM, Thompson MJ, Wellwood I, Abel GA, Hamilton W, Johnson M, Lyratzopoulos G, Messenger MP, Neal RD, Rubin G, Singh H, Spencer A, Sutton S, Vedsted P, Emery JD. Evaluating diagnostic strategies for early detection of cancer: the CanTest framework. BMC Cancer. 2019 Jun 14;19(1):586. doi: 10.1186/s12885-019-5746-6. PMID 31200676
- [Background] Murphy DR, Giardina TD, Satterly T, Sittig DF, Singh H. An Exploration of Barriers, Facilitators, and Suggestions for Improving Electronic Health Record Inbox-Related Usability: A Qualitative Analysis. JAMA Netw Open. 2019 Oct 2;2(10):e1912638. doi: 10.1001/jamanetworkopen.2019.12638. PMID 31584683
- [Background] Gandhi TK, Singh H. Reducing the Risk of Diagnostic Error in the COVID-19 Era. J Hosp Med. 2020 Jun;15(6):363-366. doi: 10.12788/jhm.3461. No abstract available. PMID 32490798
- [Background] Giardina TD, Royse KE, Khanna A, Haskell H, Hallisy J, Southwick F, Singh H. Health Care Provider Factors Associated with Patient-Reported Adverse Events and Harm. Jt Comm J Qual Patient Saf. 2020 May;46(5):282-290. doi: 10.1016/j.jcjq.2020.02.004. Epub 2020 Feb 21. PMID 32362355
- [Background] Cifra CL, Dukes KC, Ayres BS, Calomino KA, Herwaldt LA, Singh H, Reisinger HS. Referral communication for pediatric intensive care unit admission and the diagnosis of critically ill children: A pilot ethnography. J Crit Care. 2021 Jun;63:246-249. doi: 10.1016/j.jcrc.2020.09.011. Epub 2020 Sep 18. PMID 32980235
- [Background] Zimolzak AJ, Shahid U, Giardina TD, Memon SA, Mushtaq U, Zubkoff L, Murphy DR, Bradford A, Singh H. Why Test Results Are Still Getting "Lost" to Follow-up: a Qualitative Study of Implementation Gaps. J Gen Intern Med. 2022 Jan;37(1):137-144. doi: 10.1007/s11606-021-06772-y. Epub 2021 Apr 27. PMID 33907982
- [Background] Meyer AND, Giardina TD, Khawaja L, Singh H. Patient and clinician experiences of uncertainty in the diagnostic process: Current understanding and future directions. Patient Educ Couns. 2021 Nov;104(11):2606-2615. doi: 10.1016/j.pec.2021.07.028. Epub 2021 Jul 15. PMID 34312032
- [Background] Vaghani V, Wei L, Mushtaq U, Sittig DF, Bradford A, Singh H. Validation of an electronic trigger to measure missed diagnosis of stroke in emergency departments. J Am Med Inform Assoc. 2021 Sep 18;28(10):2202-2211. doi: 10.1093/jamia/ocab121. PMID 34279630
- [Background] Murphy DR, Savoy A, Satterly T, Sittig DF, Singh H. Dashboards for visual display of patient safety data: a systematic review. BMJ Health Care Inform. 2021 Oct;28(1):e100437. doi: 10.1136/bmjhci-2021-100437. PMID 34615664
- [Background] Sittig DF, Lakhani P, Singh H. Applying requisite imagination to safeguard electronic health record transitions. J Am Med Inform Assoc. 2022 Apr 13;29(5):1014-1018. doi: 10.1093/jamia/ocab291. PMID 35022741
- [Background] Sittig DF, Sengstack P, Singh H. Guidelines for US Hospitals and Clinicians on Assessment of Electronic Health Record Safety Using SAFER Guides. JAMA. 2022 Feb 22;327(8):719-720. doi: 10.1001/jama.2022.0085. No abstract available. PMID 35129591
- [Background] Singh H, Connor DM, Dhaliwal G. Five strategies for clinicians to advance diagnostic excellence. BMJ. 2022 Feb 16;376:e068044. doi: 10.1136/bmj-2021-068044. No abstract available. PMID 35172968
- [Background] Shafer GJ, Singh H, Thomas EJ, Thammasitboon S, Gautham KS. Frequency of diagnostic errors in the neonatal intensive care unit: a retrospective cohort study. J Perinatol. 2022 Oct;42(10):1312-1318. doi: 10.1038/s41372-022-01359-9. Epub 2022 Mar 4. PMID 35246625
- [Background] Giardina TD, Choi DT, Upadhyay DK, Korukonda S, Scott TM, Spitzmueller C, Schuerch C, Torretti D, Singh H. Inviting patients to identify diagnostic concerns through structured evaluation of their online visit notes. J Am Med Inform Assoc. 2022 May 11;29(6):1091-1100. doi: 10.1093/jamia/ocac036. PMID 35348688
- [Background] Shen L, Levie A, Singh H, Murray K, Desai S. Harnessing Event Report Data to Identify Diagnostic Error During the COVID-19 Pandemic. Jt Comm J Qual Patient Saf. 2022 Feb;48(2):71-80. doi: 10.1016/j.jcjq.2021.10.002. Epub 2021 Oct 29. PMID 34844874
- [Background] Read AJ, Waljee AK, Sussman JB, Singh H, Chen GY, Vijan S, Saini SD. Testing Practices, Interpretation, and Diagnostic Evaluation of Iron Deficiency Anemia by US Primary Care Physicians. JAMA Netw Open. 2021 Oct 1;4(10):e2127827. doi: 10.1001/jamanetworkopen.2021.27827. PMID 34596670
- [Background] Sittig DF, Singh H. Policies to Promote Shared Responsibility for Safer Electronic Health Records. JAMA. 2021 Oct 19;326(15):1477-1478. doi: 10.1001/jama.2021.13945. No abstract available. PMID 34505867
- [Background] Zhou Y, Walter FM, Mounce L, Abel GA, Singh H, Hamilton W, Stewart GD, Lyratzopoulos G. Identifying opportunities for timely diagnosis of bladder and renal cancer via abnormal blood tests: a longitudinal linked data study. Br J Gen Pract. 2021 Dec 31;72(714):e19-e25. doi: 10.3399/BJGP.2021.0282. Print 2022 Jan. PMID 34903517
- [Background] Bradford A, Shahid U, Schiff GD, Graber ML, Marinez A, DiStabile P, Timashenka A, Jalal H, Brady PJ, Singh H. Development and Usability Testing of the Agency for Healthcare Research and Quality Common Formats to Capture Diagnostic Safety Events. J Patient Saf. 2022 Sep 1;18(6):521-525. doi: 10.1097/PTS.0000000000001006. Epub 2022 Apr 22. PMID 35443253
- [Background] Ramesh S, Ayres B, Eyck PT, Dawson JD, Reisinger HS, Singh H, Herwaldt LA, Cifra CL. Impact of subspecialty consultations on diagnosis in the pediatric intensive care unit. Diagnosis (Berl). 2022 Apr 11;9(3):379-384. doi: 10.1515/dx-2021-0137. eCollection 2022 Aug 1. PMID 35393849
- [Background] Giardina TD, Hunte H, Hill MA, Heimlich SL, Singh H, Smith KM. Defining Diagnostic Error: A Scoping Review to Assess the Impact of the National Academies' Report Improving Diagnosis in Health Care. J Patient Saf. 2022 Dec 1;18(8):770-778. doi: 10.1097/PTS.0000000000000999. Epub 2022 Apr 27. PMID 35405723
- [Background] Meyer AND, Scott TMT, Singh H. Adherence to National Guidelines for Timeliness of Test Results Communication to Patients in the Veterans Affairs Health Care System. JAMA Netw Open. 2022 Apr 1;5(4):e228568. doi: 10.1001/jamanetworkopen.2022.8568. PMID 35452111
- [Background] Fischer H, Hahn EE, Li BH, Munoz-Plaza CE, Luong TQ, Harrison TN, Slezak JM, Sim JJ, Mittman BS, Lee EA, Singh H, Kanter MH, Reynolds K, Danforth KN. Potentially Harmful Medication Dispenses After a Fall or Hip Fracture: A Mixed Methods Study of a Commonly Used Quality Measure. Jt Comm J Qual Patient Saf. 2022 Apr;48(4):222-232. doi: 10.1016/j.jcjq.2022.01.003. Epub 2022 Jan 13. PMID 35190249
- [Background] Makris KI, Clark DL, Buffie AW, Steen EH, Ramsey DJ, Singh H. Missed Opportunities to Promptly Diagnose and Treat Adrenal Tumors. J Surg Res. 2022 Aug;276:174-181. doi: 10.1016/j.jss.2022.02.049. Epub 2022 Mar 30. PMID 35366423
- [Background] Cifra CL, Tigges CR, Miller SL, Curl N, Monson CD, Dukes KC, Reisinger HS, Pennathur PR, Sittig DF, Singh H. Reporting Outcomes of Pediatric Intensive Care Unit Patients to Referring Physicians via an Electronic Health Record-Based Feedback System. Appl Clin Inform. 2022 Mar;13(2):495-503. doi: 10.1055/s-0042-1748147. Epub 2022 May 11. PMID 35545126
- [Background] Bradford A, Shofer M, Singh H. Measure Dx: Implementing pathways to discover and learn from diagnostic errors. Int J Qual Health Care. 2022 Sep 10;34(3):mzac068. doi: 10.1093/intqhc/mzac068. PMID 36047352
- [Background] Bradford A, Singh H. Building clinical pathways of the future that improve safety and reduce waste in healthcare. J Hosp Med. 2023 Feb;18(2):200-201. doi: 10.1002/jhm.13044. Epub 2023 Jan 12. No abstract available. PMID 36633160
- [Derived] Zubkoff L, Zimolzak AJ, Meyer AND, Sloane J, Shahid U, Giardina T, Memon SA, Scott TM, Murphy DR, Singh H. A Virtual Breakthrough Series Collaborative for Missed Test Results: A Stepped-Wedge Cluster-Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2440269. doi: 10.1001/jamanetworkopen.2024.40269. PMID 39476237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Records from VA's Data warehouse (Fecal Occult Blood Test, Hep C Virus, Mammogram, alpha feto protein, dual energy x-ray absorptiometry, human papillomavirus, Chest X-ray, and Chest CT) Medical records suspicious for breast, lung, bladder, hepatocellular, and colorectal cancer.
  All data collected at the site level; number enrolled reflects number of sites enrolled
  Michael E. DeBakey VA Medical Center, Houston, Texas White River Junction VA Medical Center, White River Junction, Vermont
Pre-assignment Details: Exclusion criteria:
  Medical records that don't contain any tests, procedures, or appointments that need to be followed up on.
Units Other Than Participants: Sites
Groups:
- Sequence 1: 7 months of pre intervention, 6 months of action phase, 13 months of continuous improvement
- Sequence 2: 14 months of pre intervention, 6 months of action phase, 6 months of continuous improvement
- Sequence 3: 20 months of pre intervention, 6 months of action phase
Period: Pre Intervention for All Sites
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected)
Completed | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Not Completed | NA; 0 Sites | NA; 0 Sites | NA; 1 Sites
Period: Action Phase for Sequence 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Completed | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Not Completed | NA; 0 Sites | NA; 0 Sites | NA; 0 Sites
Period: Action Phase for Sequence 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Completed | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Not Completed | NA; 0 Sites | NA; 0 Sites | NA; 0 Sites
Period: Action Phase for Sequence 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Completed | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 4 Sites (Participant level data were not collected; only data at the site level were collected) | NA; 3 Sites (Participant level data were not collected; only data at the site level were collected)
Not Completed | NA; 0 Sites | NA; 0 Sites | NA; 0 Sites

BASELINE CHARACTERISTICS:
Population: Participant level data were not collected; only data at the site level were collected
Units Other Than Participants: Sites
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 4 | 4 | 3 | 11
Number analyzed (Sites) | 4 | 4 | 3 | 11
Age, Customized [Count of Units; unit: Sites] — Data on the baseline measures for Age, Customized" and "Sex/Gender, Customized were not collected Population: Participant level data were not collected; only data at the site level were collected
  Sites
    number analyzed (Participants) | 0 | 0 | 0 | 0
    Not Reported | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Units; unit: Sites] — Data on the baseline measures for Age, Customized" and "Sex/Gender, Customized were not collected
  Sites
    Not Reported | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    (all) |  |  |  | 0
Region of Enrollment [Number; unit: participants] — Population: Participant level data were not collected; only data at the site level were collected
  participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    United States : Northeast | 2 | 0 | 2 | 4
    United States : West | 1 | 1 | 0 | 2
    United States : Midwest | 0 | 2 | 0 | 2
    United States : South | 1 | 1 | 1 | 3
Percentage of abnormal test results with timely follow-up action [Number; unit: percentage] — Baseline data are collected from each site in the stepped-wedge trial before contact with the study team
  Reporting measure type: Percentage of tests with timely follow-up across all sites. Population: Participant level data were not collected; only data at the site level were collected
  percentage
    number analyzed (Participants) | 0 | 0 | 0 | 0
    Baseline percentage for lung follow up | 65.1 | 73.3 | 77.4 | 72.1
    Baseline percentage for Fecal Occult Blood Test follow up | 77.1 | 72.1 | 80.4 | 75.9

OUTCOME MEASURES:

1. Primary Outcome: Trigger Outcome
Description: Percentage of missed test results determined by electronic indicators. The percentage of test results with timely follow up was calculated for each participating site, out of all abnormal tests at that site.
  Reporting measure type: Percentage of tests with timely follow-up across all sites.
Time Frame: 32 months
Measure: Number; unit: percentage of abnormal tests w/ followup
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 4 | 4 | 3
percentage of abnormal tests w/ followup
  percent abnormal chest imaging tests with follow up | 67.0 | 65.9 | 78.6
  percent abnormal Fecal Occult Blood tests with follow up | 78.1 | 67.7 | 78.2

2. Primary Outcome: External Peer Review Program (EPRP) Outcome
Description: Percentage of patients notified of actionable test results within seven days via EPRP
Time Frame: 32 months
Population: Data could not be reported because EPRP measures are aggregated quarterly. Our previous understanding was that these data was granular enough for the needed breakdown of data by month. On final analysis, however, the action phases did not align with EPRP quarters, so EPRP rates could not be assigned correctly to action phase vs other phases.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 32 months
Description: Adverse events were assessed at site level and not participant level. No adverse events were reported.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04166240/Prot_SAP_000.pdf